CLINICAL TRIAL: NCT05637684
Title: Influence of Low Intensity Pulsed Ultrasound on Enhancing Biostimulation of Median Nerve in Patients With Chronic Carpal Tunnel Syndrome
Brief Title: Low Intensity Ultrasound in Patients With Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, fahd abdelazim hassan abdelgalil, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LIPUS
Record Dates: First submitted 2022-11-14; First posted 2022-12-05 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low intensity pulsed ultrasound group (Experimental): low intensity pulsed ultrasound application The following parameters will be used: intensity of 0.3 W/cm2 at a 1megahertz frequency for 20 minutes and pulsed (20%) ultrasound waves and conventional physical therapy program will be used for this group in a form of wrist hand Splint ,Medical Massage (effleurage),Passive stretching for wrist flexor, Carpal mobilization and Strengthening exercise
  Interventions: Device: low intensity pulsed ultrasound
- control group (Sham Comparator): conventional physical therapy program will be used for this group in a form of wrist hand Splint ,Medical Massage (effleurage),Passive stretching for wrist flexor, Carpal mobilization and Strengthening exercise
  Interventions: Device: low intensity pulsed ultrasound

INTERVENTIONS:
Device: low intensity pulsed ultrasound — mechanical sound waves

SUMMARY:
To investigate the influence of low intensity pulsed ultrasound on Pain level, pinch grip strength, sensory distal latency of the median nerve, motor distal latency of the median nerve and hand function in patients with chronic carpal tunnel syndrome

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) is an entrapment neuropathy caused by compression of the median nerve as it travels through the wrist's carpal tunnel. It is the most common nerve entrapment neuropathy, accounting for 90% of all neuropathies. Early symptoms of carpal tunnel syndrome include pain, numbness, and paresthesia. These symptoms typically present, with some variability, in the thumb, index finger, middle finger, and the radial half (thumb side) of the ring finger. Pain also can radiate up the affected arm. With further progression, hand weakness, decreased fine motor coordination, clumsiness, and thenar atrophy can occur.

Low-intensity ultrasound (LIU) and low-intensity pulsed ultrasound (LIPUS) are known to have positive effects on dentin genesis, cell proliferation, protein synthesis, collagen synthesis, membrane permeability, and integrin expression and to increase cytosolic calcium levels.

ELIGIBILITY:
Inclusion Criteria:

1. 26 male and 26 female patients have unilateral with mild to moderate CTS in dominant hand diagnosed and referred by physician.
2. Age will be ranged from 30-50 years
3. All patients have body mass index between 18.5 and 24.9 kg/m2
4. Median nerve sensory distal latency > 3.5 millisecond but not more than 4.5 millisecond, motor distal latency longer than 4.2 millisecond but not exceed 6.5 millisecond.
5. Positive clinical manifestation (pain, paresthesia in the distribution of the median nerve for 6 months, positive Tinel's and Phalen's sign)

Exclusion Criteria:

1. Patients with diabetes mellitus ( type I or type II),
2. Patients with hypothyroidism
3. Patients with rheumatoid disease
4. Patients with renal disease
5. Patients with polyneuropathy
6. patients with cervical radiculopathy
7. Patients with wrist arthritis , wrist fracture and acute trauma
8. Patients with Carpal tunnel release surgery
9. Patients with outlet syndrome
10. thenar muscle atrophy -

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
median nerve sensory distal latency | 4 WEEKS
  Measurements of sensory distal latency of median nerve (Antidromic technique )
  1. Recording electrode or Ring electrode (R1, R2): at the index finger the negative electrode is between 2-3 cm to positive electrode (Distance between stimulating and recording sites 5 cm).
  2. Stimulating site (S): at the wrist (Middle of the wrist between the tendons to the flexor carpi radialis and palmaris longus) Ground (Earth) electrode (G): between stimulating and recording electrodes will be placed at the palmar surface of the wrist crease.
median nerve motor distal latency | 4 WEEKS
  Measurements of motor distal latency of median nerve (Using Orthodromic technique)
  1. Recording (-) active electrode (R1): abductor pollicis brevis (APB). Reference(+) electrode (R2): placed over the first metacarpal-phalangeal joint
  2. Stimulating electrode (S): 2 stimulating sites at wrist and antecubital fossa (Cathode toward recording electrode).
  3. Ground (Earth) electrode (G): around the wrist crease between stimulating and recording electrodes
pinch grip strength | 4 weeks
  grip strength will be measured using a calibrated baseline hydraulic dynamometer, while the subject will be seated with the arm adducted, elbow flexed at 90 degree, forearm in neutral position firstly, therapist will ask patient to hold the dynamometer between the tip of the thumb and tip of the index finger it called (tip to tip pinch), as hard as possible in the hand to be tested, the patients strongly encouraged to give a maximum effort. One practice trial, Repeat the test 3 times and calculate an average with one min rest in between

CONTACTS AND LOCATIONS:
Overall Officials: FAHD A HASSAN, Principal Investigator — Cairo University
Locations (1):
- Faculty of Physical Therapy Cairo University, Giza, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: No